CLINICAL TRIAL: NCT01651195
Title: Probiotic and Respiratory and Gastrointestinal Tract Infections in Finnish Military Conscripts - a Randomized and Placebo-controlled Double-blinded Study
Brief Title: Probiotics and Infections in Conscripts in Military Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Finnish Defense Forces (Other Government); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Anne pitkäranta, Professor/Chief Physician at Hospital District of Helsinki and Uusimaa, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 189/13/03/00/11
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Tract Infections; Gastrointestinal Diseases; Asthma Exacerbations
MeSH Terms: conditions — Respiratory Tract Infections; Gastrointestinal Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotic tablet (military recruits) (Active Comparator): Lactobacillus rhamnosus 8-9 x 10 -9 2 x 2 3 weeks
  Interventions: Dietary Supplement: Probiotic; Other: Placebo
- Placebo tablet (military recruits) (Placebo Comparator): Crystalline cellulose 2 x 2, 3 weeks
  Interventions: Dietary Supplement: Probiotic; Other: Placebo
- Probiotic tablet (reserve officer candidates) (Active Comparator): Lactobacillus rhamnosus 8-9 x 10 -9 2 x 2 3 weeks
  Interventions: Dietary Supplement: Probiotic; Other: Placebo
- Placebo tablet (reserve officer candidates) (Placebo Comparator): Crystalline cellulose 2 x 2, 3 weeks
  Interventions: Dietary Supplement: Probiotic; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
Other: Placebo

SUMMARY:
The aim was to study whether probiotic intervention has an impact on seasonal occurrence of upper respiratory and gastrointestinal infections in two different conscript groups. In a randomised, double-blinded, placebo controlled study a total of 983 healthy adults were enrolled from two intakes of conscripts. Conscripts were randomised to receive either a probiotic combination of Lactobacillus rhamnosus GG (LGG) and Bifidobacterium animalis ssp. lactis BB12 (BB12) or a control chewing tablet twice daily for 150 days (recruits) or for 90 days (reserve officer candidates). Clinical examinations were carried out and daily symptom diaries were collected. Outcome measures were the number of days with respiratory and gastrointestinal symptoms and symptom incidence, number and duration of infection episodes, number of antibiotic treatments received and number of days out of service because of the infection. Statistically no significant differences were found between the intervention groups either in the risk of symptom incidence or duration. However, probiotic intervention was associated with reduction of specific respiratory infection symptoms in military recruits, but not in reserve officer candidates. Probiotics did not significantly reduce overall respiratory and gastrointestinal infection morbidity.

DETAILED DESCRIPTION:
Military conscripts are susceptible to respiratory and gastrointestinal tract infections. In previous studies probiotics have shown potency to reduce upper respiratory and gastrointestinal infections. The aim was to study whether probiotic intervention has an impact on seasonal occurrence of upper respiratory and gastrointestinal infections in two different conscript groups. In a randomised, double-blinded, placebo controlled study a total of 983 healthy adults were enrolled from two intakes of conscripts. Conscripts were randomised to receive either a probiotic combination of Lactobacillus rhamnosus GG (LGG) and Bifidobacterium animalis ssp. lactis BB12 (BB12) or a control chewing tablet twice daily for 150 days (recruits) or for 90 days (reserve officer candidates). Clinical examinations were carried out and daily symptom diaries were collected. Outcome measures were the number of days with respiratory and gastrointestinal symptoms and symptom incidence, number and duration of infection episodes, number of antibiotic treatments received and number of days out of service because of the infection. Statistically no significant differences were found between the intervention groups either in the risk of symptom incidence or duration. However, probiotic intervention was associated with reduction of specific respiratory infection symptoms in military recruits, but not in reserve officer candidates. Probiotics did not significantly reduce overall respiratory and gastrointestinal infection morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults attending military service in July 2012 and healthy adults attending reserve office school in October 2012

Exclusion Criteria:

* Regular use of oral corticosteroids
* Regular consumption (over 3 times a week) of probiotic bacteria containing products 3 weeks before intervention

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 983 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne I Pitkäranta, md, Principal Investigator — Chief Physician
Locations (2):
- Finland (2):
  - The Finnish Defence Forces, Hamina
  - The Finnish Defence Forces, Upinniemi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalima K, Lehtoranta L, He L, Pitkaniemi J, Lundell R, Julkunen I, Roivainen M, Narkio M, Makela MJ, Siitonen S, Korpela R, Pitkaranta A. Probiotics and respiratory and gastrointestinal tract infections in Finnish military conscripts - a randomised placebo-controlled double-blinded study. Benef Microbes. 2016 Sep;7(4):463-71. doi: 10.3920/BM2015.0172. Epub 2016 Apr 6. PMID 27048835

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sample size was calculated on the assumption that the use of probiotic would result in a 17% reduction in the number of sick days estimated that, with a power of 85% and at a significance level of 0.05 (Power 0.85, ß=0.15000 and α=0.05), we needed 300 conscripts per group to show a 17% difference between the groups. Each conscript was randomly allocated to the probiotic or the control group according to a computer generated, 8-blocked randomization list.
Groups:
- Probiotic Tablet (Military Recruits); Probiotic Tablet (Reserve Officer Candidates): Lactobacillus rhamnosus 8-9 x 10 -9 2 x 2 3 weeks
  Probiotic
- Placebo Tablet (Military Recruits); Placebo Tablet (Reserve Officer Candidates): Chrystalline celluloce 2 x 2, 3 weeks
  Placebo
Period: Overall Study
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
Started | 284 | 284 | 204 | 211
Completed | 63 | 73 | 121 | 103
Not Completed | 221 | 211 | 83 | 108

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates) | Total
Number analyzed (Participants) | 284 | 284 | 204 | 211 | 983
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 284 | 284 | 204 | 211 | 983
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 284 | 284 | 204 | 211 | 983
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 284 | 284 | 204 | 211 | 983

OUTCOME MEASURES:

1. Primary Outcome: Number of Sick Days
Description: The number of sick days with respiratory and gastrointestinal symptoms and symptom incidence. Other outcome measures were the number and duration of infection episodes, the number of antibiotic treatments received, and the number of days out of service due to an infection. Respiratory infection episodes and symptomatic days were counted by the basis of respiratory infection symptoms recorded into the symptom diary and from the medical visits to health care centers. If the conscript showed minimum of two RTI symptoms for a period of one day or one RTI symptom for a period of two days a RTI episode was considered to be present. Between two episodes a minimum of seven days of non-symptomatic period should be experienced if to be considered as two separate infections. If there were less non-symptomatic days, it was considered to be a continuation of the same infection episode. Symptomatic days were days when at least one symptom was experienced.
Time Frame: Through study completion, an average of 4 months
Population: According to the study nurse, the file containing number of sick days data of this particular study is no more available.
Units Other Than Participants: Days
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
Number analyzed (Participants) | 0 | 0 | 0 | 0
Number analyzed (Days) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Probiotic Tablet (Military Recruits) vs Placebo Tablet (Military Recruits) vs Probiotic Tablet (Reserve Officer Candidates) vs Placebo Tablet (Reserve Officer Candidates); Test type: Superiority — We estimated that, with a power of 85% and at a significance level of 0.05 (Power 0.85, ß=0.14990 and α=0.05), we needed 467 conscripts per group to show a 17% difference between the groups. Each conscript was randomly allocated to the probiotic or the control group according to a computer generated, 8-blocked randomization list; p < 0.05, Fisher Exact; Result variables were analyzed according to "intention to treat" (ITT) principle. Missing data was handled by statistic modeling. Data on symptom diaries were calculated as follows: the incidence and duration of individual infection symptoms and respiratory episodes were analyzed between the intervention groups using time to event analysis (cox model for hazard) and duration analysis (gamma regression model). The results are expressed as a hazard ratio (incidence rate ratio) of symptoms and the mean duration of symptoms (days) with 95% confidence intervals or standard deviations. The sums of respiratory and gastrointestinal symptoms were calculated with gamma regression analysis

2. Secondary Outcome: Number and Duration of Infection Episodes
Description: Respiratory infection episodes and symptomatic days were counted by the basis of respiratory infection symptoms recorded into the symptom diary and from the medical visits to health care centers.
Time Frame: Through study completion, an average of 4 months
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Groups:
- Placebo Tablet (Military Recruits); Placebo Tablet (Reserve Officer Candidates): Crystalline cellulose 2 x 2, 3 weeks
  Placebo
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
Number analyzed (Participants) | 284 | 284 | 204 | 211
Number analyzed (Episodes) | 411 | 402 | 56 | 101
Episodes | 33 | 35 | 30 | 29
Statistical Analysis 1: Comparison: Probiotic Tablet (Military Recruits) vs Placebo Tablet (Military Recruits) vs Probiotic Tablet (Reserve Officer Candidates) vs Placebo Tablet (Reserve Officer Candidates); Test type: Superiority; p < 0.05, Fisher Exact

3. Secondary Outcome: Number of Antibiotic Treatments Received
Description: Number of antibiotic treatments received were collected during the medical visits.
Time Frame: Through study completion, an average of 4 months
Measure: Count of Units; unit: Treatments
Units Other Than Participants: Treatments
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
Number analyzed (Participants) | 284 | 284 | 204 | 211
Number analyzed (Treatments) | 91 | 88 | 17 | 31
Treatments | 15 | 23 | 2 | 1
Statistical Analysis 1: Comparison: Probiotic Tablet (Military Recruits) vs Placebo Tablet (Military Recruits) vs Probiotic Tablet (Reserve Officer Candidates) vs Placebo Tablet (Reserve Officer Candidates); Test type: Superiority; p < 0.05, Fisher Exact

4. Secondary Outcome: Number of Days Out of Service Due to an Infection
Description: If the conscript showed minimum of two RTI symptoms for a period of one day or one RTI symptom for a period of two days a RTI episode was considered to be present. Between two episodes a minimum of seven days of non-symptomatic period should be experienced if to be considered as two separate infections. If there were less non-symptomatic days, it was considered to be a continuation of the same infection episode. Symptomatic days were days when at least one symptom was experienced. Gastrointestinal tract infection episodes and symptom days were calculated in the same fashion except 14 non symptomatic days should be in between the two to be considered as two different episodes.
Time Frame: Through study completion, an average of 4 months
Measure: Count of Units; unit: Days
Units Other Than Participants: Days
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
Number analyzed (Participants) | 284 | 284 | 204 | 211
Number analyzed (Days) | 150 | 150 | 90 | 90
Days | 44 | 41 | 4 | 6
Statistical Analysis 1: Comparison: Probiotic Tablet (Military Recruits) vs Placebo Tablet (Military Recruits) vs Probiotic Tablet (Reserve Officer Candidates) vs Placebo Tablet (Reserve Officer Candidates); Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Probiotic Tablet (Military Recruits) | Placebo Tablet (Military Recruits) | Probiotic Tablet (Reserve Officer Candidates) | Placebo Tablet (Reserve Officer Candidates)
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/284 | 0/204 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/284 | 0/204 | 0/211
Other Adverse Events (participants affected / at risk) | 0/284 | 0/284 | 0/204 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No